CLINICAL TRIAL: NCT00445796
Title: Randomised, Comparative Study of the Efficacy and Safety of Arsucam® Administered as a Single Daily Intake Versus Two Daily Intakes in the Treatment of Plasmodium Falciparum Malaria Attack
Brief Title: Arsucam® (Artesunate + Amiodaquine) Efficacy and TOLerance
Acronym: ATOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0163
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artesunate; Amodiaquine

INTERVENTIONS:
Drug: Artesunate
Drug: Amodiaquine

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority, in terms of clinical and parasitological efficacy on Day 14, of administration of Arsucam® as a single daily intake versus two daily intakes.

Secondary Objective:

To compare the clinical safety of the two treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* weighing ≥ 10 kg
* residing in the area covered by the investigating centre throughout the entire follow-up period
* axillary temperature ≥ 37.5 degrees Celsius or history of fever within the previous 24 hours
* Plasmodium falciparum density in the blood ranging from 1000 to 100,000 asexual forms per cubic millimetre

Exclusion Criteria:

* presence of at least one sign of severe malaria or clinical danger sign : prostration, consciousness disorders, recent and repeated convulsions , respiratory distress, inability to drink, uncontrollable vomiting, macroscopic haemoglobinuria, jaundice, haemorrhagic shock, systolic Blood Pressure < 70 mmHg in adults or < 50 in children, spontaneous bleeding, inability to sit or stand
* serious concomitant disease
* allergy to one of the investigational medicinal products
* pregnant women or breast-feeding women.
* documented intake of an antimalarial at a suitable dosage within seven days prior to inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2005-06

PRIMARY OUTCOMES:
clinical and parasitological cure on Day 14
Secondary: incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Lameyre, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis, Yaoundé, Cameroon
- Sanofi-Aventis, Dakar, Senegal